CLINICAL TRIAL: NCT06798207
Title: A Phase 2 Clinical Trial of TQB2102 for Injection in the Treatment of Patients With Recurrent/Metastatic Advanced Gynecological Tumors to Evaluate the Safety and Efficacy
Brief Title: A Clinical Trial of TQB2102 for Injection in Gynecological Tumors With Recurrent/Metastatic Advanced
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-II-05
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-12

CONDITIONS: Gynecological Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2102 for injection (Experimental): Intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle
  Interventions: Drug: TQB2102 for injection

INTERVENTIONS:
Drug: TQB2102 for injection — TQB2102 for injection is a HER2 dual-antibody-drug Conjugate (ADC).

SUMMARY:
TQB2102 is an antibody-drug conjugate comprised of a humanised antibody against Human Epidermal Growth Factor Receptor 2 (HER2), a enzyme-cleavable linker, and a topoisomerase I inhibitor payload, which combine the ability of antibodies to specifically target tumour cells with the highly potent killing activity of drugs with payloads too toxic for systemic administration. This is a Phase 2 study to evaluate the efficacy,and safety of TQB2102 for injection in recurrent/metastatic advanced gynecological tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study, sign informed consent and have good compliance.
* The age is ≥ 18 years old (subject to the date of signing the informed consent); Female ; eastern cooperative oncology group (ECOG ) score 0-1 ; estimated survival time ≥ 3 months ;
* Histologically confirmed, unresectable recurrent / metastatic advanced gynecologic tumors;
* The HER2 expression status (IHC 3+, 2+, 1+ or 0) is confirmed in the tumor tissue, and the subjects with completely negative IHC 0 staining are excluded.
* Previous chemotherapy with platinum-based drugs was unsuccessful.
* There is at least one measurable lesion according to the RECIST 1.1 criteria; women of childbearing potential need to meet the following conditions: the serum/urine pregnancy test result is negative before the first administration; they agree to adopt highly effective contraceptive measures (with an annual failure rate of less than 1%) throughout the study period. Women of childbearing potential are defined as premenopausal women who have not had a record of tubal ligation or hysterectomy, or women who have been postmenopausal for no more than 1 year.

Exclusion Criteria:

* Other malignant tumors occurred within the past 5 years before treatment or currently suffered simultaneously.
* Uncontrollable toxic reactions above CTCAE Grade 1 caused by any previous treatment, excluding alopecia.
* Received major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days before the start of treatment.
* Long-term unhealed wounds or fractures.
* Subjects with a history of interstitial lung disease/pneumonia ( non-infectious type ) that required steroid drug intervention treatment in the past, or currently accompanied by interstitial lung disease/pneumonia, or those with suspected interstitial lung disease/pneumonia indicated by screening imaging and cannot be excluded.
* Subjects with moderate to severe pulmonary dysfunction/disease within 3 months before the first administration.
* Arterial/deep vein thrombosis events occurred within 6 months before treatment, such as cerebrovascular accidents, deep vein thrombosis, and pulmonary embolism.
* Subjects with any severe and/or uncontrolled diseases.
* Patients with local recurrence suitable for surgery or radiotherapy.
* Those with disease progression after receiving chemotherapy drugs of topoisomerase I inhibitors or ADC drugs with small molecule toxins as topoisomerase I inhibitors in the previous first-line treatment.
* Any anti-cancer therapy or any other experimental drug treatment within 28 days or 5 half-lives before the first administration in this study.
* Received treatment with Chinese patent medicines with clear anti-tumor indications in the drug instructions approved by National Medical Products Administration (NMPA) within 2 weeks before the first administration in this study.
* Serosal effusion that requires repeated drainage to relieve clinical symptoms, or those who received serosal effusion drainage for treatment purposes within 2 weeks before treatment.
* Patients with clinically significant tumor bleeding or perforation within 1 month before the start of the study treatment, or any bleeding event ≥ CTCAE Grade 3, or patients with bleeding or coagulation disorders who are using warfarin, aspirin, or other antiplatelet aggregation drugs.
* Subjects with known central nervous system metastasis and/or carcinomatous meningitis, with diffuse dissemination. Subjects with a history of brain metastasis may be considered for inclusion if clinically stable.
* Severe bone damage and spinal cord compression caused by tumor bone metastasis, including weight-bearing bone pathological fractures that occurred within 6 months or are likely to occur in the near future, poorly controlled severe bone pain, etc.
* Those allergic to macromolecular drug components or allergic to any research drug, any component or excipient in the drug.
* Received live attenuated vaccines within 4 weeks before treatment.
* Active autoimmune diseases that required systemic treatment (such as using disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the first administration.
* Received systemic glucocorticoid treatment or any other form of immunosuppressive therapy or diagnosed with immunodeficiency within 2 weeks before treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Baseline up to 12 months
  ORR defined as percentage of participants achieving complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Duration of remission (DOR) | Baseline up to 12 months
  DOR defined as the time when the participants first achieved complete or partial remission to disease progression.
Progression-free survival (PFS) | Baseline up to 12 months
  PFS defined as the time from the first injection until the first documented progressive disease (PD) or death from any cause, whichever happens first.
Overall survival (OS) | Baseline up to 17 months
  OS defined as the time from the first injection to death from any cause.
Disease control rate (DCR) | Baseline up to 12 months
  DCR defined as percentage of participants achieving complete response (CR), partial response (PR) and stable disease (SD).
Frequency of adverse event (AE) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first
  The occurrence of all adverse medical events after the first injection.
Severity of adverse event (AE) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The severity of all adverse medical events after the first injection.
Anti-drug antibody (ADA) | Before infusion on cycle1 day1, cycle2 day1,cycle 4 day1, cycle7 day1, cycle12 day1 (each cycle is 21 days), 30 days after the end of the last infusion
  Incidence of anti-drug antibody (ADA).

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Cancer Hospital Chinise Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Maternal and Child Health Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - GanSu Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Meizhou peoples Hospital, Meizhou, Guangdong
  - Affiliated Qingyuan Hospital, Guangzhou Medical University,Qingyuan People's Hospital, Qingyuan, Guangdong
  - Affiliated Qingyuan Hospital,Guangzhou Medical University,Qingyuan People's Hospital, Qingyuan, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hostipal, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Ruijin Hospital, Shanghai Jiaotong University School of Med, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer center, Shanghai, Shanghai Municipality
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Second Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Affiliated Cancer Hospital, Ürümqi, Xinjiang
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang